CLINICAL TRIAL: NCT03077828
Title: Phase II Trial of Pembrolizumab in Combination With ICE Salvage Chemotherapy for Relapsed/Refractory Hodgkin Lymphoma
Brief Title: Pembrolizumab and Combination Chemotherapy in Treating Patients With Relapsed or Refractory Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jane N. Winter, Jane N. Winter, M.D., Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 16H07; NU 16H07 (Other: Northwestern University); P30CA060553 (NIH); NCI-2016-01439 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00203658 (Other: Northwestern University IRB#)
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Results first posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Lymphocyte-Rich Classical Hodgkin Lymphoma; Recurrent Lymphocyte-Depleted Classical Hodgkin Lymphoma; Recurrent Mixed Cellularity Classical Hodgkin Lymphoma; Recurrent Nodular Sclerosis Classical Hodgkin Lymphoma; Refractory Lymphocyte-Depleted Classical Hodgkin Lymphoma; Refractory Mixed Cellularity Classical Hodgkin Lymphoma; Refractory Nodular Sclerosis Classical Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Carboplatin; Etoposide; Ifosfamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, etoposide, carboplatin, ifosfamide) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1, etoposide IV over 60 minutes on days 1-3 of courses 1-2, carboplatin IV over 60 minutes on day 2 of courses 1-2, and ifosfamide IV over 24 hours on day 2 of courses 1-2. Pembrolizumab in combination with ICE chemotherapy repeats every 21 days for 2 courses, patients will then receive pembrolizumab as monotherapy on course 3.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
The purpose of this research study is to evaluate a new drug Pembrolizumab in combination with chemotherapy, for Relapsed/Refractory Hodgkin Lymphoma. The chemotherapy regimen is called "ICE" and includes three drugs: ifosfamide, carboplatin, and etoposide. Pembrolizumab is currently Food and Drug Administration (FDA) approved for the treatment of some patients with melanoma, lung cancer and head and neck cancer, but has not yet been approved for the treatment of Relapsed/Refractory Hodgkin Lymphoma. The 'ICE' regimen of chemotherapy is currently FDA approved for the treatment of Relapsed/Refractory Hodgkin Lymphoma, but has not yet been investigated in combination with pembrolizumab for this disease. For patients who have a relapse of their Hodgkin's lymphoma, retreatment with chemotherapy followed by a stem cell transplant is recommended. We know that obtaining a complete remission (not able to detect any disease on scans) is very important prior to proceeding to the stem cell transplant. Patients with negative scans have a lower chance of the disease coming back and a higher chance of achieving a long-term cure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete response rate by fludeoxyglucose- positron emission tomography/computed tomography (FDG-PET/CT) prior to autologous hematopoietic stem cell transplant (AHSCT) with the combination of pembrolizumab and ifosfamide, carboplatin, etoposide (ICE) salvage chemotherapy for relapsed/refractory Hodgkin lymphoma.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of pembrolizumab in combination with salvage high-dose chemotherapy according to Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.03.

II. To estimate the event free survival (EFS) at 2 years from start of treatment.

III. To estimate the overall survival (OS) at 2 years from start of treatment.

TERTIARY OBJECTIVES:

I. To characterize PD-1 pathway specific expression and correlate with response.

II. To characterize serum biomarkers of immune and inflammatory response during treatment.

III. To characterize levels of soluble PD-L1 related to treatment with pembrolizumab.

IV. To characterize T-lymphocyte subset changes to treatment with pembrolizumab.

V. To investigate the prevalence and clinical correlation of chromosome 9p24.1 mutations for this population.

VI. To evaluate the effect on stem cell harvest following treatment with pembrolizumab.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1, etoposide IV over 60 minutes on days 1-3 of courses 1-2, carboplatin IV over 60 minutes on day 2 of courses 1-2, and ifosfamide IV over 24 hours on day 2 of courses 1-2. Pembrolizumab in combination with ICE chemotherapy repeats every 21 days for 2 courses, patients will then receive pembrolizumab as monotherapy on course 3.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of classical Hodgkin lymphoma including nodular sclerosis, mixed cellularity, lymphocytic-rich, and lymphocyte depleted subtypes by the 4th edition of the World Health Organization (WHO) Classification of Tumors of Hematopoietic and Lymphoid Tissues published in 2008
* Patients must have disease with FDG-PET/CT avidity
* Patients must have relapsed/refractory disease, with at least one line of prior chemotherapy, but =< 2 prior lines of treatment, for Hodgkin lymphoma; NOTE: Patients must not have had prior immune checkpoint inhibitors; however, there are no other limitations to prior agent or regimen types
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Patients must have adequate organ and bone marrow function within 10 days of registration, as defined below:
* Absolute neutrophil count >= 1,000/mcL (in the absence of granulocyte colony stimulating factor (GCSF) for >= 14 days)
* Platelets >= 75,000/mcl (in the absence of platelet transfusion for >= 14 days)
* Hemoglobin >= 7g/dL (transfusion permitted)
* Total bilirubin =< 2 x institutional upper limit of normal (ULN); if total bilirubin is > 2 x ULN, the direct bilirubin must be normal
* Aspartate aminotransferases (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SPGT]) =< 2.5 x institutional ULN
* Creatinine =< 2 x ULN or creatinine clearance (CrCl) > 30 ml/min
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to registration; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Females of childbearing potential (FOCBP) should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy
  * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months) NOTE: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy, monoclonal antibody (mAb), or targeted small molecule therapy within 4 weeks of study registration are not eligible; those who have not recovered from adverse events (grade 1 or baseline) due to such agents administered more than 4 weeks earlier are not eligible
* Patients may not be currently receiving any other investigational agents within 4 weeks of study registration
* Patients must not have had prior exposure to any immune checkpoint inhibitors including anti-PD-1, anti-PD-L1 agents, anti-PD-L2 agents, or anti-CTLA-4 monoclonal antibodies
* Patients must not have known central nervous system (CNS) involvement
* Patients must not have had prior stem cell transplantation (autologous or allogeneic)
* Patients must not have persistent diarrhea greater than National Cancer Institute (NCI) CTCAE grade 2 at the time of study registration, despite medical management
* Patients must not have a history of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, noninfectious pneumonitis
* Patients with known immunodeficiency, known autoimmune disease, or concurrent use of immunomodulatory agents including systemic steroids within 7 days prior to registration, are ineligible
* Patients must not have co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens; this includes, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not have a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Patients with known human immunodeficiency virus (HIV) infection or active TB (Bacillus tuberculosis) are not eligible
* Patients with known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection are not eligible
* Patients must not have a hypersensitivity to pembrolizumab or any of its excipients
* Patients must not have received a live vaccine within 30 days of registration Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed)
* Patients must not be pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Patients who are unwilling or unable to comply with the protocol or have known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2024-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jane N. Winter, M.D., Principal Investigator — Northwestern University
Locations (6):
- United States (6):
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Rochester, Rochester, New York

REFERENCES:
- [Derived] Bryan LJ, Casulo C, Allen PB, Smith SE, Savas H, Dillehay GL, Karmali R, Pro B, Kane KL, Bazzi LA, Chmiel JS, Palmer BA, Mehta J, Gordon LI, Winter JN. Pembrolizumab Added to Ifosfamide, Carboplatin, and Etoposide Chemotherapy for Relapsed or Refractory Classic Hodgkin Lymphoma: A Multi-institutional Phase 2 Investigator-Initiated Nonrandomized Clinical Trial. JAMA Oncol. 2023 May 1;9(5):683-691. doi: 10.1001/jamaoncol.2022.7975. PMID 36928527

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient started treatment 04/24/2017. The study was designed to enroll patients with relapsed/refractory classical Hodgkin lymphoma following standard up-front chemotherapy. The study was closed to further enrollment on 10/29/2020 due to meeting accrual goal.
Groups:
- Treatment: Patients received treatment with combination pembrolizumab and ICE (ifosphamide, carboplatin, etoposide) salvage chemotherapy for 2 cycles (1 cycle = 21 days). Pembrolizumab 200 mg IV will be administered on day 1. Standard ICE salvage chemotherapy includes ifosfamide 5 g/m2 with equivalent dose of MESNA given over 24 hours by CIV on day 2, carboplatin AUC 5 IV with a maximum of 800 mg on day 2, and etoposide 100 mg/m^2/day IV on days 1 to 3. G-CSF support administered 24 hours following completion of chemotherapy.
  On Cycle 3 day1, patients received pembrolizumab monotherapy. An FDG-PET/CT will be obtained 14-22 days after pembrolizumab monotherapy to assess response by Deauville criteria. Patients with Deauville </= 3 will proceed to AHSCT which may include a 4th optional cycle of Pembro-ICE prior to transplant per investigator discretion. Patients with Deauville >3 will be treated per provider's discretion which may also include stem cell transplant.
Period: Treatment Cycles
Arm/Group | Treatment
Started | 43
Cycle 1 | 42
Cycle 2 | 39
Cycle 3 | 39
Optional Cycle 4 (Cycle #4 is not required on the study protocol. Patients with a Deauville score ≤3 may proceed directly to AHSCT per provider discretion if the procedure can be arranged within 21-35 days after cycle #3. Alternatively, if the patient's FDG-PET/CT has a Deauville score >3, they will come off protocol, receive no further study agent, and be treated per investigator discretion.) | 5
Completed | 39
Not Completed | 4
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Screen Fail | 2
Period: Autologous Stem Cell Transplant
Arm/Group | Treatment
Started (Autologous Stem Cell Transplant will took place 21-42 days after the final study regimen pembrolizumab dose (optional pembro-ICE combination or otherwise, per provider discretion). Transplant visit parameters were obtained on the initial day of induction chemotherapy or within 21-42 days following final study regimen but prior to the autologous stem cell transplant procedure.) | 42
Completed | 38
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1
Period: Follow-up
Arm/Group | Treatment
Started | 39
Completed | 24
Not Completed | 15
Not completed — Patients still in follow-up | 15

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 32
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: To determine the complete response rate by FDG-PET/CT prior to AHSCT with the combination of pembrolizumab and ICE salvage chemotherapy for relapsed/refractory Hodgkin lymphoma. Response was assessed using Lugano criteria 2014.
  To address the primary aim, the proportion of patients with complete responses was calculated(defined as FDG-PET/CT Deauville score ≤ 3) as (number of responders) / (number of evaluable patients).
Time Frame: Up to 59 days
Population: Of the 42 registered study patients, 37 were evaluable for response.
  To be evaluable for inclusion in the analysis to address the primary objective, patients must:
  * have received at least dose of pembrolizumab AND
  * have a FDG-PET/CT scan following cycle #3
Measure: Count of Participants; unit: Participants
Groups:
- Treatment: Patients receive pembrolizumab IV over 30 minutes on day 1, etoposide IV over 60 minutes on days 1-3 of courses 1-2, carboplatin IV over 60 minutes on day 2 of courses 1-2, and ifosfamide IV over 24 hours on day 2 of courses 1-2. Pembrolizumab in combination with ICE chemotherapy repeats every 21 days for 2 courses, patients will then receive pembrolizumab as monotherapy on course 3.
  Carboplatin: Given IV
  Etoposide: Given IV
  Ifosfamide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
Arm/Group | Treatment
Number analyzed (Participants) | 37
Participants
  Complete Repsonse | 32
  Partial Response | 4
  Progressive Disease | 1

2. Secondary Outcome: Incidence of Adverse Events
Description: Evaluate the safety and tolerability of pembrolizumab in combination with ICE salvage high-dose chemotherapy by measuring the frequency and severity of adverse events by type, severity (grade), timing, and attribution to pembrolizumab which will be assessed according the NCI-CTCAE version 4.03.
Time Frame: Up to 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Event Free Survival (EFS)
Description: EFS will be defined as the length of time from treatment on protocol until the first occurrence of disease relapse, progression, re-initiation of cytotoxic chemotherapy, or death due to disease, or until last contact if the patient did not experience any of these, assessed up to 2 years.
Time Frame: Up to 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival (OS)
Description: OS will be defined as time from study enrollment until death, or until last contact if the patient did not die, assessed up to 2 years.
Time Frame: Up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All adverse events were monitored and recorded from the time of consent for up to four cycles of treatment,( 1 Cycle = 21 days) during stem-cell transplant ( up to 42 days after the last cycle) and up to 180 days post stem-cell transplant.
Description: Data collected includes the highest grade of the event experienced for each participant, and thus includes some serious adverse event data.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 1/42
Serious Adverse Events (participants affected / at risk) | 17/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=42)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Fever (General disorders) | 2
Lymphocyte count decreased (Blood and lymphatic system disorders) | 2
Platelet count decrease (Blood and lymphatic system disorders) | 2
Sepsis (Infections and infestations) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Ejection fraction decrease (Cardiac disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hematoma (Vascular disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Infusion related reaction (General disorders) | 1
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1
Engraftment syndrome (Investigations) | 1
Mucositis Oral (Gastrointestinal disorders) | 1
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1
Pericardial tamponade (Cardiac disorders) | 1
Respiratory failure (Reproductive system and breast disorders) | 1
Skin infection (Skin and subcutaneous tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=42)
Anemia (Blood and lymphatic system disorders) | 41
Lymphocyte count decrease (Blood and lymphatic system disorders) | 41
Platelet count decrease (Blood and lymphatic system disorders) | 41
White blood cell decreased (Blood and lymphatic system disorders) | 40
Neutrophil count decreased (Blood and lymphatic system disorders) | 38
Nausea (Gastrointestinal disorders) | 35
Aspartate aminotransferase increased (Investigations) | 33
Hypoalbuminemia (Metabolism and nutrition disorders) | 33
Hypokalemia (Metabolism and nutrition disorders) | 33
Alanine aminotransferase increased (Investigations) | 32
Hyperglycemia (Metabolism and nutrition disorders) | 31
Hypocalcemia (Metabolism and nutrition disorders) | 31
Alkaline phosphatase increased (Investigations) | 29
Diarrhea (Gastrointestinal disorders) | 29
Hypophosphatemia (Metabolism and nutrition disorders) | 24
Hypertension (Respiratory, thoracic and mediastinal disorders) | 23
Vomiting (Gastrointestinal disorders) | 22
Constipation (Gastrointestinal disorders) | 21
Fever (General disorders) | 21
Hyponatremia (Metabolism and nutrition disorders) | 20
Mucositis oral (Gastrointestinal disorders) | 20
Fatigue (General disorders) | 17
Headache (Nervous system disorders) | 16
Alopecia (Skin and subcutaneous tissue disorders) | 15
Hypotension (Vascular disorders) | 15
Abdominal pain (Gastrointestinal disorders) | 14
Insomnia (Psychiatric disorders) | 14
Hypomagnesemia (Metabolism and nutrition disorders) | 13
Maculopapular rash (Skin and subcutaneous tissue disorders) | 13
Anorexia (Metabolism and nutrition disorders) | 12
Febrile neutropenia (Blood and lymphatic system disorders) | 12
Pain (General disorders) | 12
Sinus tachycardia (Cardiac disorders) | 12
Sore throat (Respiratory, thoracic and mediastinal disorders) | 12
Gastroesophageal reflux disease (Gastrointestinal disorders) | 11
Chills (General disorders) | 10
Anxiety (Psychiatric disorders) | 9
Dizziness (Nervous system disorders) | 9
Dry mouth (Gastrointestinal disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Weight loss (Metabolism and nutrition disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Creatinine increased (Investigations) | 7
Esophagitis (Gastrointestinal disorders) | 7
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 7
Infections and infestations - Other (Infections and infestations) | 7
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 6
Oral Pain (Gastrointestinal disorders) | 6
Sepsis (Infections and infestations) | 6
Blood bilirubin increase (Investigations) | 5
Edema limbs (General disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
General disorders and administration site conditions - Other (General disorders) | 5
Hot flashes (Vascular disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 5
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 5
Sinus bradycardia (Cardiac disorders) | 5
Bloating (Gastrointestinal disorders) | 4
Cardiac disorders - Other (Cardiac disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 4
Depression (Psychiatric disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 4
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4
Localized edema (General disorders) | 4
Lung infection (Infections and infestations) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
pain in extremity (Musculoskeletal and connective tissue disorders) | 4
radiation recall reaction (dermtologic) (Injury, poisoning and procedural complications) | 4
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4
Skin infection (Skin and subcutaneous tissue disorders) | 4
Dysgeusia (Nervous system disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 3
Lethargy (Nervous system disorders) | 3
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Renal and urinary disorders - Other (Renal and urinary disorders) | 3
Syncope (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 3
Urinary tract infection (Renal and urinary disorders) | 3
Vascular access complication (Injury, poisoning and procedural complications) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT03077828/Prot_SAP_000.pdf